CLINICAL TRIAL: NCT04437290
Title: University of Washington Alzheimer's Disease Research Center (UW ADRC) Imaging & Biomarker Core
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Ellison Foundation (Unknown)
Responsible Party: Principal Investigator, Thomas Grabowski, Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00009617; P30AG066509 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer Disease
Keywords: mild cognitive impairment; dementia; tau
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer disease: The group is composed of individuals with a consensus diagnosis of amnestic mild cognitive impairment (MCI) or amnestic multimodal MCI or dementia primarily attributed to Alzheimer's disease (AD), as determined by the UW ADRC Clinical Core. They will have age of presentation > 55 years, sporadic onset, CDR (Clinical Dementia Rating Scale) score 0.5-1.0, and sufficient English competency to complete a standardized cognitive testing battery. All will have no contraindication to MRI and will have had an MRI scan in the UW ADRC Imaging and Biomarker Core. These participants will undergo PET scanning with the investigational tau tracer [18F] MK6240
  Interventions: Drug: investigational radiotracer [18F]MK6240

INTERVENTIONS:
Drug: investigational radiotracer [18F]MK6240 — Brain PET scan

SUMMARY:
This is a cross-sectional, observational study that characterizes research participants with Alzheimer's disease (AD) for their patterns of brain degeneration with the investigational tau positron emission tomography (PET) radiotracer [18F] MK-6240. The goal is to describe the topographic pattern of involvement of cerebral brain regions (topographic phenotyping) in early stage AD participants using tau PET in a sub-cohort of the University of Washington Alzheimer's Disease Research Center (ADRC) Clinical Cohort, and to make this phenotype information available to affiliated research studies at the University of Washington and to the general scientific community via the National Alzheimer's Coordinating Center.

DETAILED DESCRIPTION:
Memory loss and dementia, including Alzheimer's disease (AD), are heterogeneous in terms of pattern of symptoms and brain atrophy, likely due to underlying variability in AD biological processes, as well as comorbidity (separate diseases that co-occur with AD). The correspondence between clinical findings and underlying cause is imperfect, though, and the field has benefitted tremendously from development of biomarkers that can be used for diagnosis, for estimation of the biological burden of pathology, and/or for tracking disease trajectories. For example, in the National Institute on Aging-Alzheimer's Association (NIA-AA) research framework, biomarkers of Amyloid beta, phosphorylated Tau, and Neurodegeneration (A/T/N) standardize the separation of cases with Alzheimer pathophysiology from those without it.

A sub-cohort of UW ADRC Clinical Core participants who have amyloid deposition (A+ by cerebrospinal fluid [CSF] or amyloid PET) and mild degrees of cognitive impairment will be investigated for their specific pattern of tau deposition with tau PET. Additionally, participants who are thought to be resilient to Alzheimer disease, e.g. 85 years or older and normal cognition, or A+ by CSF or amyloid PET and normal cognition, will also be investigated for their specific pattern of tau deposition with tau PET.

The ADRC Imaging and Biomarker Core will conduct and analyze these scans, and store the data in the Integrated Brain Imaging Center at the University of Washington Medical Center campus, which is directed by the PI, Dr. Grabowski. It will also use other data collected by ADRC Cores (such as neuropsychology testing) to perform other analysis, such as estimating resilience measures (i.e. the ability of the brain to function well in spite of the presence of AD).

This sub-cohort will aid in the investigation of Alzheimer's disease and related dementias (ADRD) by providing a means to better understand the relationships between the spatial patterns of tau deposition, neurodegeneration in the brain, cognitive symptoms, and resilience. It will provide a ready source of potential participants to the larger research community. By standardizing and supporting the collection imaging and CSF for research participants with Alzheimer's disease and related dementias under the ADRC, we promote research synergism and productivity across UW studies of AD and related disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Amnestic MCI or Amnestic multimodal MCI or dementia primarily attributed to AD, by consensus diagnosis in the ADRC Clinical Core;
2. Evidence of A+ T+ Alzheimer disease by CSF evaluation (e.g. low amyloid beta(AB)42 or 42/40 ratio and elevated p-181-tau); or evidence of A+ Alzheimer disease by amyloid PET.
3. Age of presentation for first evaluation > 55 years;
4. Sporadic onset, defined by not from a known autosomal dominant AD family and not more than 1 first degree relative with dementia onset before age 65;
5. Clinical Dementia Rating scale (CDR) score 0.5 or 1.0;
6. English competency sufficient to complete cognitive testing battery to the satisfaction of ADRC neuropsychologist;
7. MRI scan in the Clinical Core, with additional selection for topographic diversity, based on the MRI imaging.

Exclusion Criteria:

1. History of symptomatic cerebrovascular disease (CVD) or CVD evaluated to contribute significantly to cognitive impairments;
2. Parkinsonism, or meeting revised McKeith criteria for possible or probable Dementia with Lewy bodies;
3. Contraindication to MRI scanning (e.g. metal implants, severe claustrophobia);
4. Premorbid history of neurologic disease that may contribute to cognitive impairment (e.g. multiple sclerosis, epilepsy, brain tumor);
5. History of developmental dyslexia or other developmental disorder affecting validity of cognitive tests. These exclusion criteria minimize comorbidity;
6. Pregnancy or breast-feeding.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with preclinical, prodromal, or mild dementia due to Alzheimer's disease, based on amyloid biomarker evidence
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
tau PET SUVR image | Day 1
  Parametric [18F]MK6240 standardized uptake ratio images (SUVR) generated using an inferior cerebellar gray matter reference region.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Grabowski, MD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified tau PET scans will be shared with the National Alzheimer's Coordinating Center (NACC) through the Standardized and Centralized Alzheimer's Neuroimaging initiative (U24), which will make these data available under a data use agreement to non-commercial entities and non- commercial research projects.
  De-identified tau PET scans will be shared with Cerveau Technologies, Inc, for their own Imaging Core database of tau PET scans internationally, under terms of our Master Research Agreement. Non-identifying information about the participants, e.g. age, sex, apolipoprotein E (APOE) genotype, research diagnosis, is also to be included in the Cerveau imaging core database.
Supporting Information: Study Protocol, CSR
Time Frame: tau PET imaging data will be uploaded to NACC within 6 months of data acquisition.
  tau PET imaging data will be uploaded to Cerveau Technologies, Inc within 6 months of data acquisition
Access Criteria: per National Alzheimer's Coordinating Center policy
  per Cerveau Technologies, Inc policy
URL: http://www.alz.washington.edu

REFERENCES:
- [Background] Lohith TG, Bennacef I, Vandenberghe R, Vandenbulcke M, Salinas CA, Declercq R, Reynders T, Telan-Choing NF, Riffel K, Celen S, Serdons K, Bormans G, Tsai K, Walji A, Hostetler ED, Evelhoch JL, Van Laere K, Forman M, Stoch A, Sur C, Struyk A. Brain Imaging of Alzheimer Dementia Patients and Elderly Controls with 18F-MK-6240, a PET Tracer Targeting Neurofibrillary Tangles. J Nucl Med. 2019 Jan;60(1):107-114. doi: 10.2967/jnumed.118.208215. Epub 2018 Jun 7. PMID 29880509
- [Background] Pascoal TA, Shin M, Kang MS, Chamoun M, Chartrand D, Mathotaarachchi S, Bennacef I, Therriault J, Ng KP, Hopewell R, Bouhachi R, Hsiao HH, Benedet AL, Soucy JP, Massarweh G, Gauthier S, Rosa-Neto P. In vivo quantification of neurofibrillary tangles with [18F]MK-6240. Alzheimers Res Ther. 2018 Jul 31;10(1):74. doi: 10.1186/s13195-018-0402-y. PMID 30064520
- [Background] Koole M, Lohith TG, Valentine JL, Bennacef I, Declercq R, Reynders T, Riffel K, Celen S, Serdons K, Bormans G, Ferry-Martin S, Laroque P, Walji A, Hostetler ED, Briscoe RJ, de Hoon J, Sur C, Van Laere K, Struyk A. Preclinical Safety Evaluation and Human Dosimetry of [18F]MK-6240, a Novel PET Tracer for Imaging Neurofibrillary Tangles. Mol Imaging Biol. 2020 Feb;22(1):173-180. doi: 10.1007/s11307-019-01367-w. PMID 31111397